CLINICAL TRIAL: NCT00881036
Title: Activation of HBV Under Immunosuppression in HBsAg-negative But Anti-HBc-positive Patients With Hematological Malignancies
Brief Title: Activation of Hepatitis B Virus (HBV) in Hepatitis B Surface Antigen (HBsAg) - Negative But Hepatitis B Core Antibody (Anti-HBc) - Positive Patients
Status: Completed | Type: Observational
Sponsor: Kyoto University (Other)
Responsible Party: Principal Investigator, Yoshihide Ueda, Associate Professor, Kyoto University
Organization: Kyoto University Hospital (Other)
Other Study IDs: HBV from anti-HBc positive
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis B
Keywords: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Individuals with resolved hepatitis B, characterized as hepatitis B surface antigen (HBsAg)-negative and hepatitis B core antibody-positive, have latent hepatitis B virus (HBV) infection in their liver tissue. Cytotoxic chemotherapy and hematopoietic stem cell transplantation sometimes trigger the reactivation of latently infected HBV, resulting in de novo hepatitis B. Although de novo hepatitis B could cause acute liver failure or chronic hepatitis, an effective management strategy for de novo hepatitis B has not been well established. Risk factors and effective management for de novo hepatitis B will be clarified.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg-negative but anti-HBc-positive

Exclusion Criteria:

* Serum HBV DNA-negative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBsAg-negative but anti-HBc-positive patients with hematological malignancies treated at Kyoto University Hospital
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2006-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kyoto Univesity, Kyoto, Kyoto, Japan